CLINICAL TRIAL: NCT00712270
Title: A Randomized Double-blind Trial of Aripiprazole and Risperidone in Schizophrenia: An Evaluation of Neuroimaging, Neuropsychological, and Pharmacogenomic Markers of Differential Treatment Response
Brief Title: Best Event Schizophrenia Trial--A Randomized Double-Blind Trial of Aripiprazole and Risperidone in Schizophrenia
Acronym: BEST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to failure to meet sufficient enrollment for valid analysis
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-009
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2018-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic drug treatment response; Risperidone; Aripiprazole; Fallypride; Positron emission tomography; Magnetic Resonance Imaging; Dopamine D2 Receptors
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (No Intervention): Screening and Baseline Procedures followed by Referral to Community Care. Baseline Procedures may be repeated at a later time if appropriate.
- Drug: Aripiprazole (Active Comparator): Screening and Baseline Procedures followed by 16 weeks of treatment with aripiprazole, followed by repeat of baseline procedures and referral to community care.
  Interventions: Drug: Aripiprazole
- Risperidone (Active Comparator): Screening and Baseline Procedures followed by 16 weeks of treatment with Risperidone,followed by repeat of baseline procedures and referral to community care.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Aripiprazole — Target dose = 15mg by mouth per day for 16 weeks. The dosage will be titrated in accordance with the treating physician's clinical judgment, generally reaching full dosage within one week of initiation. The dosage may be increased as clinically indicated, by the treating physician. Any deviation from these target dosing schedules must be reviewed and approved by the principal investigator, generally prior to the adjustment unless clinical circumstances require more immediate adjustment (in which case the treating physician should consult with the principal investigator as soon as is practically possible).
  Other Names: Abilify
  Arms: Drug: Aripiprazole
Drug: Risperidone — Target Dose = 2mg by mouth per day for 16 weeks. The dosage will be titrated in accordance with the treating physician's clinical judgment, generally reaching full dosage within one week of initiation. The dosage may be increased as clinically indicated, by the treating physician. Any deviation from these target dosing schedules must be reviewed and approved by the principal investigator, generally prior to the adjustment unless clinical circumstances require more immediate adjustment (in which case the treating physician should consult with the principal investigator as soon as is practically possible).
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
This study is being conducted to find a way to predict how individual schizophrenic patients will respond if they are treated with different types of antipsychotic drugs. This could help doctors prescribe the medication that will work best for each individual.

DETAILED DESCRIPTION:
The primary objective of the proposed research project is to identify a practical method of predicting differential antipsychotic drug treatment response in patients with schizophrenia. In particular, we will examine differential response to two antipsychotic drugs, aripiprazole and risperidone, that have contrasting pharmacologic activity at D2-type dopamine receptors, i.e., partial agonism vs. antagonism, respectively. A number of candidate predictors will be examined, including neuroimaging parameters (regional neuroanatomical and metabolic variations, fallypride binding to D2-like receptors), neuropsychological testing, clinical features, laboratory measures, and genetic studies.

Secondary objectives include: (1) extension of our previous efforts to characterize abnormalities in cortico-striato-thalamic circuits in unmedicated schizophrenics using PET and MR imaging; and, (2) examination of the role of omega-3 fatty acid activity in schizophrenics as a predictor of dopaminergic activity.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will meet DSM-IV diagnostic criteria for schizophreniform disorder, schizophrenia, schizoaffective disorder or (non-affective) psychotic disorder, NOS. Subjects with schizophreniform disorder or psychotic disorder, NOS, will be diagnostically reevaluated (recontacted if no longer involved in the study) after a minimum of six months of psychotic symptoms in order to determine whether diagnostic criteria for schizophrenia or schizoaffective disorder have been met.
2. Subjects will be between 18 and 55 years of age, inclusive.
3. Subjects will be able to fully participate in the informed consent process, or have a legal guardian able to participate in the informed consent process.
4. Present score on at least one PANSS psychosis items (P1, P2, P3, P5 or P6) > 4(moderately severe) and CGI Severity score > 4 (moderate).
5. Female patients of childbearing potential must be using a medically accepted means of contraception

Exclusion Criteria:

1. Current active substance use disorder diagnosis or a history of cocaine abuse or dependence;
2. Female patients who are either pregnant or nursing;
3. Known history of mental retardation, seizure disorder, or a clinically significant head injury (prolonged loss of consciousness, neurological sequelae, or demonstrated structural brain injury);
4. Non-English speaking (mastery of English insufficient to participate in study evaluation procedures);
5. Serious, unstable medical illness;
6. Known hypersensitivity to any study medication;
7. Medical contraindication to any element of the study procedure;
8. Current symptoms which present serious risk of danger to self or others;
9. Participation in a clinical trial of an investigational drug within 30 days of study entry;
10. Current severity of psychiatric symptoms contraindicates a delay in initiation of antipsychotic medication treatment until functional imaging studies and neuropsychological testing have been completed;
11. Baseline QTc interval of > 450 msec.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Lehrer, MD, Principal Investigator — Wallace Kettering Neuroscience Institute
Locations (1):
- Wallace Kettering Neuroscience Institute, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Entire Study Population: The study was pre-maturely terminated and limited data is available for reporting, since none of the study team members currently work in the organization, and are not able to be contacted. The randomization coding is not available, therefore, results cannot be reported per-Arm.
Period: Overall Study
Arm/Group | Entire Study Population
Started (Unknown - study was terminated back in 2009 with limited data available. Randomization is not known) | 21
Completed (Unknown - study was terminated back in 2009 with limited data available. Randomization is not known) | 7
Not Completed | 14
Not completed — Withdrawal by Subject | 11
Not completed — Screen Failure | 3

BASELINE CHARACTERISTICS:
Population: The study was pre-maturely terminated and limited data is available for reporting, since none of the study team members currently work in the organization, and are not able to be contacted. No baseline data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Drug: Aripiprazole | Risperidone | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Pre and Post Treatment PET and MRI Imaging
Time Frame: At baseline and 16 weeks
Population: Study was terminated back in 2009 with limited data available. Randomization is not known. Only 7 subjects completed study. Data for this objective is not available.
Arm/Group | Standard of Care | Drug: Aripiprazole | Risperidone
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: QTc Measurement
Description: Information regarding the Outcome Measure being a Primary or Secondary, is unavailable.
Population: Limited data only available for 8 of 21 patients
Measure: Mean (Full Range); unit: milliseconds
Groups:
- QTc Pre-treatment for Entire Study Population: QTc measurement via ECG prior to treatment initiation.
- QTc Post-treat for Entire Study Population: QTc measurement via ECG after treatment initiation
Arm/Group | QTc Pre-treatment for Entire Study Population | QTc Post-treat for Entire Study Population
Number analyzed (Participants) | 8 | 8
milliseconds | 381 [350 to 412] | 389 [354 to 505]

3. Secondary Outcome: Assessment of Pretreatment and Posttreatment Psychiatric Rating Scales to Include PANSS and CGI
Description: Study was terminated back in 2009 with limited data available. Randomization is not known. Only 7 subjects completed study. Data for this objective is not available.
Time Frame: 7 visits over 16 weeks
Population: as for outcome 1
Arm/Group | Entire Study Population
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Study was terminated back in 2009 with limited data available. Randomization is not known. Only 7 subjects completed study. Data for AEs is not available.
Groups:
- Entire Study Population: Study was terminated back in 2009 with limited data available. Randomization is not known. Only 7 subjects completed study.
Arm/Group | Entire Study Population
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 14/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=21)
Decreased sexual arousal (Reproductive system and breast disorders) | 1
Increased urination (Renal and urinary disorders) | 1
Elevated serum HCG (Reproductive system and breast disorders) | 1
Post-procedure vaginal bleed (Reproductive system and breast disorders) | 1
Urinalysis abnormalities (Renal and urinary disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Delayed orgasm (Reproductive system and breast disorders) | 1
Cecal polyps (Gastrointestinal disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 1
Tooth extraction (Musculoskeletal and connective tissue disorders) | 1
Weight gain (Musculoskeletal and connective tissue disorders) | 1
Daytime sleepiness (Nervous system disorders) | 7 (7)
Akinesia (Nervous system disorders) | 4
Insomnia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 2
Akathisia (Nervous system disorders) | 1 (3)
Weakness (Musculoskeletal and connective tissue disorders) | 1
Lightheadedness (Cardiac disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 1
Dry mouth (General disorders) | 8
Sialorrhea (General disorders) | 3
Tonsilitis (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Common cold (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4 (4)
Decreased appetite (Gastrointestinal disorders) | 1
Emesis (Gastrointestinal disorders) | 1
Increased appetite (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1 (2)
GI distress (indigestion and cramping) (Gastrointestinal disorders) | 1
GERD (increased symptoms) (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Claustrophobia (General disorders) | 1 (4)
Increased sweating (Skin and subcutaneous tissue disorders) | 1
Decreased Hemoglobin and Hematocrit (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated back in 2009 with limited data available. Randomization is not known. Only 7 subjects completed study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No